CLINICAL TRIAL: NCT00720083
Title: A Randomized Phase II Trial of Chemoradiotherapy Versus Chemoradiotherapy and Vandetanib for High-Risk Postoperative Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Chemotherapy and Radiation Therapy (RT) With or Without Vandetanib in Treating Patients With High-Risk Stage III or Stage IV Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of drug supply.
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0619; CDR0000599867
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; vandetanib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT + Cisplatin (Active Comparator): Patients undergo radiotherapy 5 times a week for up to 6.5 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Radiation: radiation therapy
- RT + Cisplatin + Vandetanib (Experimental): Patients undergo radiotherapy as in arm I and receive cisplatin IV over 1 hour once a week beginning on day 1 of radiotherapy. Patients also receive oral vandetanib once daily beginning 14 days prior to the start of radiotherapy. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: vandetanib; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: vandetanib — Given orally
  Arms: RT + Cisplatin + Vandetanib
Radiation: radiation therapy — Patients undergo radiotherapy 5 times a week for up to 6.5 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving chemotherapy together with radiation therapy is more effective with or without vandetanib in treating patients with head and neck cancer.

PURPOSE: This randomized phase II trial is studying giving chemotherapy together with radiation therapy to see how well it works compared with giving chemotherapy and radiation therapy together with vandetanib in treating patients with high-risk stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To screen for an indication that the addition of vandetanib to chemoradiotherapy may prolong disease-free survival as compared to a combination of chemoradiotherapy in patients with resected, high-risk stage III or IV head and neck squamous cell carcinoma.

Secondary

* To determine whether this treatment regimen can be delivered safely and successfully following surgical resection for advanced head and neck cancer.
* To estimate the locoregional progression, distant metastasis, and overall survival rates for patients treated with this regimen.
* To examine the distribution of selected biomarkers that may include but are not limited to EGFR (epidermal growth factor receptor, total and phosphorylated), E-cadherin, pMAPK (phosphorylated mitogen-activated protein kinase), pAKT, Stat-3 (signal transducer and activator of transcription 3), Ki-67, COX-2 (cyclooxygenase 2), and cyclin B1 (G2/mitotic-specific cyclin-B1)expression in this group of patients and to explore the potential correlation between these markers with the ultimate treatment outcome

OUTLINE: This is a multicenter study. Patients are stratified according to Zubrod performance status (0 vs 1) and primary site of disease (oral cavity/hypopharynx vs larynx vs oropharynx, HPV+ (human papillomavirus positive) vs oropharynx, HPV- (human papillomavirus negative)). Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo radiotherapy 5 times a week for up to 6.5 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
* Arm II: Patients undergo radiotherapy as in arm I and receive cisplatin IV over 1 hour once a week beginning on day 1 of radiotherapy. Patients also receive oral vandetanib once daily beginning 14 days prior to the start of radiotherapy.

In both arms, treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.

Tissue samples from all patients are collected and reviewed. Tissue from patients with oropharyngeal carcinoma is analyzed for human papillomavirus.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck, including any of the following subtypes:

  * Oral cavity
  * Oropharynx
  * Larynx
  * Hypopharynx
* Stage III or IV disease (no distant metastases)
* No cancer of the lip, nasopharynx, or sinuses
* Must have undergone gross total resection* (with curative intent) within 3-6 weeks of registration, with pathology demonstrating 1 or more of the following risk factors:

  * Histologic extracapsular nodal extension
  * Invasive cancer seen on microscopic evaluation of the resection margin, when all visible tumor has been removed NOTE: *Tonsillar cancer patients who undergo transoral excision of all gross tumor are eligible if the patient has formal neck dissection confirming histologic extracapsular nodal extension

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Zubrod performance status 0-1
* ANC (absolute neutrophil count) ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention to achieve this level allowed)
* Total bilirubin normal
* AST (aspartate aminotransferase) or ALT (alanine amino transferase) ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Serum creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Glucose ≥ 40 mg/dL AND ≤ 250 mg/dL
* Sodium ≥ 130 mmol/L AND ≤ 155 mmol/L
* Magnesium ≥ 0.9 mg/dL AND ≤ 3 mg/dL (supplementation allowed)
* Potassium ≥ 4 mmol/L AND ≤ 6 mmol/L (supplementation allowed)
* Serum calcium (ionized or adjusted for albumin) ≥ 7 mg/dL AND ≤ 12.5 mg/dL (supplementation allowed)
* QTc (corrected QT interval) interval ≥ 480 msec must have 2 additional EKGs ≥ 24 hrs apart and the average QTc from the 3 screening EKGs must be < 480 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 60 days after completion of study treatment
* May not donate blood during the study or for 3 months after last dose of vandetanib

Exclusion criteria:

* Other simultaneous primary cancer
* Prior invasive malignancy (except nonmelanoma skin cancer) unless disease free for a minimum of 3 years with the exception of the following:

  * Carcinoma in situ of the cervix
  * Adequately treated basal cell or squamous cell carcinoma of the skin
  * Untreated or treated low-risk prostate cancer (defined as clinical or pathologic T1c, N0 M0, PSA (prostate-specific antigen) < 10, Gleason < 7, < 50% of the total cores positive for cancer)
* Severe, active co-morbidity, defined as follows:

  * Clinically significant cardiovascular event (e.g., myocardial infarction, superior vena cava syndrome, or New York Heart Association class II-IV) or presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia within the past 3 months
  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 3 months
  * Transmural myocardial infarction within the past 3 months
  * History of arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE [Common Terminology Criteria for Adverse Events] grade 3), or asymptomatic sustained ventricular tachycardia

    * Patients with atrial fibrillation, controlled on medication, are eligible
  * Presence of left bundle branch block
  * Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication
  * Congenital long QTc syndrome or first degree relative with unexplained sudden death under 40 years of age
  * QTc with Bazett's correction that is unmeasurable or ≥ 480 msec on screening EKG

    * Patients who are receiving a drug that has a risk of QTc prolongation are not eligible if QTc is ≥ 460 msec
  * Hypertension (systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 100 mm Hg) not controlled by medical therapy
  * Diarrhea ≥ grade 1 (increase of < 4 stools per day over baseline or mild increase in ostomy output compared to baseline)
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC (Center for Disease Control) definition (no HIV testing is required for study entry)
* Prior allergic reaction to cisplatin or vandetanib or derivatives similar to these drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy for this disease (prior chemotherapy for a different cancer allowed)
* No prior radiotherapy to the head and neck area that would result in overlap of radiotherapy fields
* More than 30 days since prior investigational agents
* More than 3 weeks since prior major surgery and recovered
* More than 2 weeks since prior and no concurrent medications that induce Torsades de Pointes
* More than 2 weeks since prior and no concurrent known potent inducers of CYP3A4 (Cytochrome P450 3A4), including rifampicin, phenytoin, carbamazepine, barbiturates, and Hypericum perforatum (St. John wort)
* No concurrent medication that may cause QTc prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Raben, MD, Principal Investigator — University of Colorado, Denver; John A. Ridge, MD, PhD, Study Chair — Fox Chase Cancer Center; Stuart J. Wong, MD, Study Chair — Medical College of Wisconsin
Locations (63):
- United States (63):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Altanta, Georgia
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Charach Cancer Center at Huron Valley - Sinai Hospital, Commerce, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Saint Elizabeth Cancer Institute at Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Memorial Sloan-Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Radiation Oncology Associates, PA, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center - Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects were registered, after which 2 did not continue to randomization due to physician preference.
Period: Overall Study
Arm/Group | RT + Cisplatin | RT + Cisplatin + Vandetanib
Started | 17 | 15
Completed | 16 (Subjects with data for the primary analysis are considered to have completed the study.) | 13
Not Completed | 1 | 2
Not completed — Ineligible | 1 | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | RT + Cisplatin | RT + Cisplatin + Vandetanib | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Median (Full Range); unit: years] | 57 [40 to 74] | 53 [39 to 76] | 57 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: This study terminated early with 34 subjects accrued out of 170 planned, therefore no analyses were performed.
Time Frame: From randomization to date of failure (local, regional, or distant progression, or death) or last follow-up. Analysis occurs after 78 failures have been reported.
Arm/Group | RT + Cisplatin | RT + Cisplatin + Vandetanib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via CTCAE (Common Terminology Criteria for Adverse Events) 3.0 then mapped to CTCAE 4.0 to report on this website. Subjects experiencing more than one of a given SAE (serious adverse event) are counted only once for that SAE. The same methodology applied for non-SAE adverse events (AE).
Groups:
- RT+ Cisplatin: Patients undergo radiotherapy 5 times a week for up to 6.5 weeks and receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | RT+ Cisplatin | RT + Cisplatin + Vandetanib
Serious Adverse Events (participants affected / at risk) | 6/16 | 4/13
Other Adverse Events (participants affected / at risk) | 16/16 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT+ Cisplatin (N=16) | RT + Cisplatin + Vandetanib (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT+ Cisplatin (N=16) | RT + Cisplatin + Vandetanib (N=13)
Anemia (Blood and lymphatic system disorders) | 9 | 1
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 5 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Blurred vision (Eye disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 6
Diarrhea (Gastrointestinal disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 13 | 10
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Dysphagia (Gastrointestinal disorders) | 13 | 11
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 13 | 10
Nausea (Gastrointestinal disorders) | 12 | 6
Oral pain (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 7 | 6
Edema face (General disorders) | 1 | 2
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 12 | 5
Fever (General disorders) | 2 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 3
Pain (General disorders) | 4 | 1
Immune system disorders - Other (Immune system disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 2 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 12 | 7
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 3 | 5
Alanine aminotransferase increased (Investigations) | 3 | 3
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 2 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 7 | 0
Platelet count decreased (Investigations) | 3 | 2
Weight loss (Investigations) | 6 | 5
White blood cell decreased (Investigations) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 9 | 6
Headache (Nervous system disorders) | 0 | 2
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 1
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 5 | 5
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study terminated early with 34 subjects accrued out of 170 planned, therefore no analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No